CLINICAL TRIAL: NCT00201357
Title: An Open, Non-Comparative Trial to Assess the Efficacy and Safety of Oral Thalidomide (THADO) in Patientswith Hormone-Refractory Prostate Cancer-A PHASE II CLINICAL TRIAL
Brief Title: An Open Trial to Assess the Efficacy and Safety of Oral Thalidomide in Patients With Hormone-Refractory Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Health Research Institutes, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T1802
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2016-03-25 (Estimated); Status verified 2016-03

CONDITIONS: Hormone-refractory Prostate Cancer
Keywords: hormone-refractory prostate cancer; thalidomide; quality of life
MeSH Terms: interventions — Thalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Thalidomide (THADO) — patients who receive thalidomide (100 mg BID).

SUMMARY:
Trial objectives: The primary objective is to determine the proportion of patients who have 50% decrease in PSA maintained for at least 4 weeks, in advanced hormone-refractory prostate cancer (HRPC) patients who receive thalidomide (100 mg BID). Secondary objectives include the objective tumor response rate for measurable lesions, the median duration of tumor response, median time to disease progression and assessments of clinical benefits, quality of life, and safety profile.

DETAILED DESCRIPTION:
* Trial objectives: The primary objective is to determine the proportion of patients who have 50% decrease in PSA maintained for at least 4 weeks, in advanced hormone-refractory prostate cancer (HRPC) patients who receive thalidomide (100 mg BID). Secondary objectives include the objective tumor response rate for measurable lesions, the median duration of tumor response, median time to disease progression and assessments of clinical benefits, quality of life, and safety profile.
* Number of patient : about 70 evaluable patients .Simon's optimal two-stage design will be used to allow early termination should sufficient evidence of non-effectiveness are collected. Thalidomide is considered non-effective if the proportion of PSA response is 14% or lower, and is worthy of further study if the proportion of response is 30% or higher. Controlling the risk for accepting thalidomide when it is non-effective to be at most 5% and the risk for rejecting thalidomide when it is effective to be at most 10%, this design calls for 26 patients at the first stage. If four or less PSA response is observed, then the study will be terminated. Otherwise, additional 44 patients will be entered at the second stage. The treatment will be rejected if a total of 14 or less PSA responses are observed out of 70 patients. This design has 70% chance of termination after the first stage if the true PSA response rate is 14% or lower. With 70 patients, the study will provide 95% assurance to claim that the difference between the estimated and true proportion will be within 11%.
* Medication and Dose: Thalidomide (THADO 50mg/cap.) 100mg, BID.
* Duration: Continue treatment until disease progression, unacceptable toxicity or when patient meets any off-study criteria.
* Efficacy assessments: % of patients with 50% decrease in PSA maintained for at least 4 weeks,Objective tumor response Median duration of tumor response Median time to disease progression, Clinical benefits pain, performance status, weight
* Quality of life (evaluated by the instruments of EORTC-QLQ-C30, FACT-prostate)Safety assessments:
* Toxicity -Adverse Event -Laboratory Test

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older.
* Histologically or cytologically confirmed adenocarcinoma of prostate that is metastatic, hormone-refractory (confirmed by testing serum testosterone), and clinically progressive following at least one prior hormonal regimen.
* Patients must have documented progression of disease on anti-androgen withdrawal, if the patient have documented progression on previous anti-androgen therapy.
* Measurable (patient with measurable bi-dimensional disease) or evaluable disease (defined as the presence of a nonmeasurable abnormality on CT or on physical examination coupled with a PSA ³ 30).
* Karnofsky performance status ³ 60%.6. Adequate bone marrow functions: Granulocyte count 1,000/mm3, Platelets 75,000/mm3, haemoglobin 8 g/dl.
* Adequate renal and liver functions: Creatinine < 1.5 mg/dl, Bilirubin < 2 mg/dl, ALT/AST less than 2.5 times the upper limit of the reference range for the institute.
* Patients with chemical or clinical hypothyroidism should have their thyroid replacement prior to starting study.
* Patients must have recovered from the effect of recent surgery (at least 4 weeks apart), radiotherapy (at least 4 weeks apart).
* Patients have ability to complete Quality of Life (QoL) questionnaires.
* Patients must sign informed consent.

Exclusion Criteria:

* Patients with advanced second primary malignancy.
* Patients with brain metastases.
* Patients with hypersensitivity to thalidomide.
* History of myocardial infarction within past 6 months, uncontrolled congestive heart failure or angina pectoris.
* Patients with orthostatic hypotension before therapy.
* Patients with NCI CTC grade 3 or greater peripheral neuropathy of any cause that is clinically detectable.
* Patients with active infection, including positive serology for HIV.
* Patients who have received chemotherapy before for treatment of metastases of prostate cancer, or received other investigational agents or corticosteroids within 4 weeks prior to enrollment of study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2002-10; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
The primary objective is to determine the proportion of patients who have 50% decrease in PSA maintained for at least 4 weeks, in advanced hormone-refractory prostate cancer (HRPC) patients who receive thalidomide (100 mg BID). | The primary objective is to determine the proportion of patients who have 50% decrease in PSA maintained for at least 4 weeks
  The primary objective is to determine the proportion of patients who have 50% decrease in PSA maintained for at least 4 weeks

SECONDARY OUTCOMES:
Secondary objectives include the objective tumor response rate for measurable lesions, the median duration of tumor response, median time to disease progression and assessments of clinical benefits, quality of life, and safety profile. | The primary objective is to determine the proportion of patients who have 50% decrease in PSA maintained for at least 4 weeks
  The primary objective is to determine the proportion of patients who have the median duration of tumor response, median time to disease progression and assessments of clinical benefits, quality of life, and safety profil

CONTACTS AND LOCATIONS:
Overall Officials: Ruey-kuen Hsieh, M.D., Principal Investigator — Taiwan cooperative oncology group
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — http://english.nhri.org.tw/inst_cancer/ca_TCOGresearch.php